CLINICAL TRIAL: NCT01007396
Title: Diagnosis of Tuberculosis Infection in Health Care Workers Using Ex-vivo Interferon-gamma Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won-Jung Koh, MD, PhD, Associated professor, school of medicine, sungkyunkwan university, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2007-09-019
Record Dates: First submitted 2009-11-02; First posted 2009-11-04 (Estimated); Results first posted 2012-01-11 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2011-12

CONDITIONS: Latent Tuberculosis Infection
Keywords: Interferon-gamma release assay
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- new healthcare workers (Other): doctors and nurses who were newly hired in 2008 at the Samsung Medical Center
  Interventions: Other: 1-step tuberculin skin test (TST) and blood sampling

INTERVENTIONS:
Other: 1-step tuberculin skin test (TST) and blood sampling — In only new healthcare workers, the 1-step TST and quantiFERON-TB Gold In-Tube test were performed.

SUMMARY:
The present study was to evaluate the usefulness of a whole-blood interferon-r release assays (IGRAs) as diagnostic tool of the latent tuberculosis infection for healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* doctors and nurses newly hired at Samsung Medical Center between February, 2008 and November, 2008.

Exclusion Criteria:

* Non-applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2008-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Won-Jung Koh, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study participants were doctors and nurses who were newly hired in 2008 at the Samsung Medical Center, a 2,000-bed referral hospital in Seoul, Korea.
Groups:
- New Healthcare Workers: a baseline 1-step tuberculin skin test (TST) and baseline QuantiFERON-TB Gold In-Tube test were performed in the new healthcare workers.
  After oner year, serial QFT-IT testing was performed for all participants, except for those who had left the hospital.
Period: Overall Study
Arm/Group | New Healthcare Workers
Started | 322
Completed | 275
Not Completed | 47
Not completed — Lost to Follow-up | 47

BASELINE CHARACTERISTICS:
Arm/Group | New Healthcare Workers
Number analyzed (Participants) | 322
Age Continuous [Median (Inter-Quartile Range); unit: years] | 24 [22 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274
  Male | 48
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 322

OUTCOME MEASURES:

1. Primary Outcome: Annual Incidence of Tuberculosis Infection Among Newly Employed Doctors and Nurses in Korea
Description: The participants performed QuaniFERON-TB Gold In-Tube test (QFT-IT test). Annual infection of tuberculosis infection was evaluated with the conversion of QFT-IT test through annual check up of QFT-IT test. The definitions for QFT-IT test conversion was based on the CDC definition (Baseline IFN-r < 0.35 IU/ml and follow-up IFN-r ≥ 0.35 IU/ml).
Time Frame: QFT-IT test was performed at enrollment and repeated at point of one year after enrollment. So, the length of timw which from the start of the first test of very first participant to the end of second test of very last participant is 2 years.
Population: Of the 322 healthcare workers (HCWs), 275 (85%) underwent repeat QuantiFERON-TB Gold In-Tube test (QFT-IT test) after 1 year of employment; the 47 participants who had resigned were excluded. Two participants with indeterminate results on the baseline QFT-IT test were excluded from the analysis.
Measure: Number; unit: number of new cases per 1000 person/year
Arm/Group | New Healthcare Workers
Number analyzed (Participants) | 273
number of new cases per 1000 person/year | 57

2. Secondary Outcome: Negative Conversion Rate in Follow-up QuantiFERON-TB Gold In-Tube Test (QFT-IT Test) After Treatment of Latent Tuberculosis Infection (LTBI)
Description: The percentage of participants with negative conversion in follow-up QFT-IT test after LTBI treatment, out of those who had QFT-IT test conversion after one year of employment and agreed to undergo treatment for LTBI according to our recommendation
  Participants with QFT-IT test conversion were recommended for LTBI therapy using 3 months of daily isoniazid and rifampicin, which was the regular treatment for LTBI in our institution.
  The QFT-IT test was repeated after LTBI therapy. Negative conversion was defined as baseline IFN-r ≥ 0.35 and follow-up IFN-r < 0.35 IU/ml.
Time Frame: 3 months after LTBI treatment
Population: Thirteen participants agreed to undergo treatment for latent tuberculosis infection and completed 3 months therapy.
Measure: Number; unit: Percentage of participants
Arm/Group | New Healthcare Workers
Number analyzed (Participants) | 13
Percentage of participants | 15

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed.
Arm/Group | New Healthcare Workers
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes